CLINICAL TRIAL: NCT00906308
Title: A Phase 3, Double-blind, Placebo-Controlled, Randomized Clinical Trial, Assessing Safety and Efficacy of MF101 for Hot Flushes and Menopausal Symptoms in Postmenopausal Women
Brief Title: A Study of MF101 in Postmenopausal Women
Acronym: HERBA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bionovo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MF-101-004
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Hot Flushes; Vasomotor Symptoms
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MF101 5 g/day (Experimental)
  Interventions: Drug: MF101 5 g/day
- MF101 10 g/day (Experimental)
  Interventions: Drug: MF101 10 g/day

INTERVENTIONS:
Drug: MF101 5 g/day — PO (orally) 5 g/day (administered twice a day, BID) for up to 12 weeks
  Arms: MF101 5 g/day
Drug: Placebo — PO (orally) matched placebo (administered twice a day, BID) for up to 12 weeks
  Arms: Placebo
Drug: MF101 10 g/day — PO (orally) 10 g/day (administered twice a day, BID) for up to 12 weeks
  Arms: MF101 10 g/day

SUMMARY:
This phase 3a study is designed to assess the safety and efficacy of MF101 on the frequency of moderate to severe hot flushes in postmenopausal women.

DETAILED DESCRIPTION:
Menopausal women often experience debilitating menopausal vasomotor symptoms and associated insomnia. Until recently, vasomotor symptoms were often treated with estrogens, which are very effective; however, randomized clinical trials have shown that postmenopausal combination hormone therapy increases the risks for stroke, cardiovascular events, and breast cancer. New, more effective, and safer treatments for menopausal vasomotor symptoms are therefore needed.

MF101, a botanical extract, is a non-hormonal investigational treatment being tested in a randomized, double-blind, placebo-controlled phase 3a clinical trial to assess the safety and efficacy of MF101 on the frequency of moderate to severe hot flushes in postmenopausal women. Approximately 1200 healthy post-menopausal women, aged 40-65, with moderate to severe hot flushes will be enrolled to determine the safety and efficacy of two doses of MF101 (5 g/day and 10 g/day) compared to placebo after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria (limited):

* Confirmed postmenopausal women aged 40-65
* Provide written informed consent

Exclusion Criteria (limited):

* History of malignancy, with the exception of certain types of skin cancer or cervical cancer
* Known carrier of BRCA1 or BRCA2
* Abnormal mammogram or breast examination suggestive of cancer within 9 months of screening
* Endometrial hyperplasia, polyps or abnormal uterine masses (with the exception of fibroids)
* Clinical evidence of active ischemic heart disease, history of cardiovascular disease, uncontrolled hypertension, or a history of transient ischemic attacks or cerebrovascular accidents
* History of deep vein thrombosis, pulmonary embolism, severe chronic diarrhea, chronic constipation, uncontrolled inflammatory bowel syndrome or disease (IBS or IBD), or unexplained weight loss
* Active liver disease or gall bladder disease
* History of chronic hepatitis B, hepatitis C, hepatitis within 3 months, or HIV infection
* Use of prescription medications or herbal/dietary supplements for the treatment of hot flushes or those with known estrogenic/progestogenic activity within required wash-out timeframes
* Use of selective receptor modulators (SERMs), aromatase inhibitors, gonadotropin-releasing hormone agonists, selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin or clonidine within required wash-out timeframes
* Chronic use of morphine or other opiates

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and efficacy of two doses of MF101 (5 g/day and 10 g/day) compared to placebo. | 12 weeks
  Safety will be measured through clinically significant findings in physical examinations, laboratory parameters, endometrial changes, abnormal uterine bleeding and any other adverse events. Efficacy will be measured by the mean change in frequency of moderate to severe hot flushes from baseline to treatment week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tagliaferri, M.D, L.Ac., Study Director — Bionovo Inc.
Locations (50):
- United States (50):
  - Arizona Research Center, Phoenix, Arizona
  - Visions Clinical Research Center, Tucson, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Northern California Research, Sacramento, California
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Compass Research, Orlando, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - OB/GYN Specialists of the Palm Beaches, West Palm Beach, Florida
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts University, Springfield, Massachusetts
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Rochester Clinical Research, Rochester, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - PMG Research, Raleigh, North Carolina
  - Hawthorne Medical Research, Winston-Salem, North Carolina
  - Rapid Medical Research, Cleveland, Ohio
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Clinical Trials of America, Eugene, Oregon
  - Advanced Clinical Research - A Division of Medford Women's Clinic, Medford, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - South Carolina Clinical Research, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - HCCA - Clinical Research Solutions, Franklin, Tennessee
  - HCCA - Clinical Research Solutions, Jackson, Tennessee
  - University of Tennessee at Memphis, Memphis, Tennessee
  - HCCA - Clinical Research Solutions, Smyrna, Tennessee
  - Benchmark Research, Austin, Texas
  - Women Partners in Health/Professional Quality Research, Austin, Texas
  - Discovery Clinical Trials, Dallas, Texas
  - R/D Clinical Research, Lake Jackson, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - University of Virginia, Charlottesville, Virginia
  - National Clinical Research, Norfolk, Virginia
  - National Clinical Research Center, Richmond, Virginia
  - Seattle Women's Health, Research and Gynecology, Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.mf101.com